CLINICAL TRIAL: NCT07142200
Title: A Clinical Study Evaluating the Efficacy and Safety of Disitamab Vedotin Combined With PD-1 Inhibitor and Radiotherapy as Bladder-preserving Therapy in Patients With Localized HER2-high Expressing Muscle-invasive Bladder Urothelial Carcinoma Following Maximal Transurethral Resection
Acronym: DECIDING
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-0409
Record Dates: First submitted 2025-07-08; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: muscle-invasive bladder cancer; Disitamab Vedotin; PD-1 Inhibitor; Radiotherapy; Bladder-preserving Therapy
MeSH Terms: conditions — Neoplasms | interventions — disitamab vedotin; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Each patient received treatment with Vediximab injection [2.0 mg/kg, Q2W, iv] and Triprolizumab injection [3mg/kg, Q2W, iv] for one cycle, followed by concurrent radiotherapy in the second cycle.
  The subjects need to undergo maximum transurethral resection of the bladder (TURBT) and imaging diagnosis, and collect urine samples before treatment. The patient will receive treatment with vediximab combined with PD-1 and radiotherapy after TURBT surgery (without the need for secondary resection).
  The subjects should receive treatment with vediximab combined with PD-1 every two weeks for a total of 12 treatment cycles, and receive radiation therapy simultaneously. The specific number of treatment cycles will be determined by the researchers based on the patient's response to the treatment and the overall condition. Patients with safety intolerance caused by any drug treatment will be reduced or discontinued according to the dosage adjustment plan specified in the protocol.
  Interventions: Drug: Disitamab Vedotin; Drug: PD-1 inhibitor; Radiation: radiotherapy

INTERVENTIONS:
Drug: Disitamab Vedotin — Each patient will receive Disitamab Vedotin injection [2.0 mg/kg, Q2W, iv], with an expected total of 12 courses of treatment. The specific number of treatment cycles is determined by researchers based on the patient's response to the treatment, tolerance to the treatment plan, and comprehensive assessment of the condition. Patients with safety intolerance caused by any drug treatment should reduce or discontinue the medication according to the dosage adjustment plan specified in the plan. The medication is diluted with physiological saline and administered intravenously for one hour.
Drug: PD-1 inhibitor — Each patient will receive Triprolizumab injection [3mg/kg, Q2W, iv], with an expected total of 12 courses of treatment. The specific number of treatment cycles is determined by researchers based on the patient's response to the treatment, tolerance to the treatment plan, and comprehensive assessment of the condition. Patients with safety intolerance caused by any drug treatment should reduce or discontinue the medication according to the dosage adjustment plan specified in the plan. The medication is diluted with physiological saline and administered intravenously for one hour.
Radiation: radiotherapy — 1. Whole bladder treatment, recommended scope of application: T2 Suggestion: The total bladder radiotherapy dose is 2Gy/day, five times a week, up to a dose of 50Gy/25 times, to cover at least 95% of the planned target volume (PTV full bladder).
     The radiation dose for shrinking the field to bladder tumors is 2Gy/day, five times a week, with a total dose of 14Gy/7 times, to cover at least 95% of the planned target dose (PTV bladder tumors).
  2. Whole pelvic radiotherapy (whole bladder+selective pelvic lymph node radiotherapy), applicable range: T3-T4a Suggestion: Whole pelvic radiotherapy at 2Gy/day, five times a week, up to a dose of 46Gy/23 times, to cover at least 95% of the planned target dose.
  Reduce the dosage to 2Gy/day for the entire bladder and up to 4Gy/twice. Bladder tumor (PTV bladder tumor) 2Gy/day, five times a week, with a total dose of 14Gy/7 times, to cover at least 95% of the planned target volume.
  The above radiotherapy plan is a suggestion, and the specific plan will

SUMMARY:
This is a prospective, open label, multicenter clinical study of vediximab combined with PD-1 and radiation therapy for bladder preservation in MIBC patients with HER-2 high expression (IHC 2+or 3+), conducted in accordance with Good Clinical Practice (GCP).

Each patient received treatment with Vediximab injection [2.0 mg/kg, Q2W, iv] and Triprolizumab injection [3mg/kg, Q2W, iv] for one cycle, followed by concurrent radiotherapy in the second cycle. Assuming a 20% improvement in the efficacy of conventional TMT bladder protection treatment, i.e. an increase in CR rate from 60% to 80%, alpha of 0.05, and beta of 0.2, a sample size of 36 is required. Considering a 20% dropout rate, 45 subjects need to be enrolled.

The subjects need to undergo maximum transurethral resection of the bladder (TURBT) and imaging diagnosis, and collect urine samples before treatment. The researchers judged that localized myometrial invasive bladder cancer with high HER2 expression could be treated with bladder conserving therapy by maximizing TURBT. The patient will receive treatment with vediximab combined with PD-1 and radiotherapy after TURBT surgery (without the need for secondary resection).

The subjects should receive treatment with vediximab combined with PD-1 every two weeks for a total of 12 treatment cycles, and receive radiation therapy simultaneously. The specific number of treatment cycles will be determined by the researchers based on the patient's response to the treatment, tolerance to the regimen, and overall judgment of the condition. Patients with safety intolerance caused by any drug treatment will be reduced or discontinued according to the dosage adjustment plan specified in the regimen.

After completing the above treatments, the pathology, imaging, and cytology of the tumor site were obtained through diagnostic TURBT or cystoscopy for tumor evaluation to assess whether complete remission was achieved. The first tumor efficacy evaluation was conducted 3 months after receiving treatment, and the researcher judged whether to continue treatment based on the patient's treatment status. After completing the treatment for the next 3 months, another tumor efficacy evaluation was conducted. After completing all 12 treatment cycles (6 months), the patient underwent two tumor evaluations at the 6th month (from the 12th month of treatment) and the 12th month (from the 24th month of treatment), respectively.

DETAILED DESCRIPTION:
MIBC has a poor prognosis, and even with radical surgery, the 5-year survival rate is less than 60%. Although immune checkpoint inhibitors have made rapid progress in the treatment of advanced bladder and urinary tract epithelial cancer in the past year, many drugs have been approved for market both domestically and internationally.

Immunosuppressants targeting PD-1 or its ligand PD-L1, including Nivolumab, Pembrolizumab, Trastuzumab, and Triprolizumab, have been proven to be a promising approach for tumor immunotherapy. The Phase III clinical trial of Pembrolizumab compared with chemotherapy for the treatment of advanced bladder and urinary tract epithelial cancer has been successful. Nivolumab has an objective efficacy rate of 24.4% in patients with advanced bladder and urinary tract epithelial cancer who have previously failed treatment. Domestic trastuzumab (targeting high PD-L1 expression) and terilelizumab have significantly improved ORR and OS in patients who have failed platinum based chemotherapy, and the DoR of beneficiary patients has been significantly prolonged. Therefore, the efficacy of anti-PD-1 monoclonal antibody in advanced bladder and urinary tract epithelial cancer has been validated. In PURE-01, Pembrolizumab achieved a complete disease response rate of 42% in preoperative neoadjuvant therapy for MIBC, greatly changing the treatment status. Terriptylimab also achieved a pCR rate of 40% in neoadjuvant therapy for MIBC.

Whether the bladder can be preserved in patients with localized MIBC has always been a hot topic in clinical research. The ANZUP 1502 study is a phase II clinical trial evaluating the combination of Pembrolizumab and concurrent chemoradiotherapy for the treatment of MIBC, with 90% of patients achieving complete remission after 24 weeks. At the same time, TMT combined with immunotherapy achieved good bladder preservation effects in both the IMMUNOPRESSE-SOGUG study (electrocautery durvalumab+Treme radiotherapy, 12 week cCR rate of 81%) and the BTCR-GU15-023 study (durvalumab+radiotherapy, cCR rate of 54.5%). Therefore, based on the excellent results of phase II clinical studies, there are currently multiple phase III clinical studies underway, including KEYNOTE-992, SWOG1806, SunRISe-2, INTACT studies, etc.

Vidiximab for injection (product code: RC48, RC48-ADC) is an innovative new therapeutic biologic developed to meet the needs of patients with HER2 expressing malignant solid tumors. The injection of vediximab mainly exerts anti-tumor effects through two pathways: one is to inhibit the activation of HER2 downstream signaling pathways (such as PI3K/AKT) by binding to HER2 molecules on the surface of tumor cells, thereby interfering with cell transcription, growth, and proliferation; The second is through the action of small molecule MMAE on microtubule proteins during mitosis, which interferes with the formation of microtubules in cells, mainly manifested as depolymerization of microtubules and induction of cell cycle arrest in the G2/M phase. RC48-C005/C09 is a combined analysis of two clinical studies, C005 and C009. The trial enrolled a total of 107 patients with advanced urothelial carcinoma who had previously received first-line or above systemic therapy but failed. Among all 107 patients, the ORR evaluated by IRC was 50.5% (95% CI: 40.6, 60.3), and the BOR evaluation results showed that 2 patients achieved CR and 52 patients achieved PR.

From a biological perspective, the combination of targeted therapy and immunotherapy can simultaneously block the HER2 signaling pathway and PD-1/PD-L1 signaling pathway, bridge PD-1 expressing T lymphocytes and HER2 expressing tumor cells, and assist T cells in recognizing and killing tumor cells. In addition, the warhead of ADC drugs can cause tumor cell destruction through cytotoxic effects (especially the destruction of microtubules by MMAE), and the release of calcitonin, heat shock proteins, and other substances on the surface of apoptotic cells can induce immunogenic cell death (ICD), thereby activating T cells. MMAE and other microtubule protein stabilizers (MSA) can directly activate antigen-presenting cells (such as dendritic cells), promote DC maturation, enhance T cell recruitment, and reduce immune suppression in tumor tissues. Therefore, the combination of anti-HER2ADC and PD-1/L1 drugs has a synergistic effect, which can improve the immunosuppressive effect in the tumor microenvironment and enhance the infiltration of immune cells into the tumor. In the RC48-C014 study, the combination of vediximab (RC48) and terilelimab (JS001) was used for mUC with previous first-line treatment failure or intolerance/unwillingness to receive cisplatin chemotherapy. The study results showed an objective response rate of 73.2%, with an objective response rate of 76% in the first-line population, including HER2 IHC (2+/3+) and PD-L1 (+); The objective response rates of HER2 IHC (2+/3+) and PD-L1 (-) patients were 75% and 87.5%, respectively. Meanwhile, there was no significant increase in treatment-related adverse reactions compared to monotherapy.

In the first phase of this study, 6 patients did not experience any DLT events within 28 days after receiving the study drug and radiotherapy. According to the definition of the first phase study, this protocol is considered safe. In the first stage of patients, the CR rate reached 83% in March, which has preliminarily returned to normal for its effectiveness. Therefore, based on the results of the first stage, further research will be conducted in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 18 years old;
* ECOG PS:0～1;
* The subjects need to undergo maximum TURBT surgery (no need for secondary resection) and imaging diagnosis. The researchers have determined that MIBC (urothelial carcinoma as the main pathological component>50%) is present, and plan to undergo radical cystectomy, lymph node dissection, and urinary diversion surgery;
* cT2-T4a N0 M0 （CT/MRI ± PET/CT）;
* Accept maximum TURBT;
* Have tissue examination specimens with TURBT;
* Expected survival period ≥ 3 months;
* The immunohistochemical staining result of the tissue after the last TURBT surgery was IHC 2+or 3+;
* The main organ function is normal (14 days before enrollment), which meets the following criteria:

  1. The standard for blood routine examination must meet the following criteria: (no blood transfusion or treatment with granulocyte colony-stimulating factor within 14 days before enrollment):

     HB≥90 g/L； ANC≥1.5×109 /L； PLT≥100×109 /L；
  2. Non functional organic diseases must meet the following criteria:

T-BIL ≤ 1.5 × ULN (upper limit of normal value); ALT and AST ≤ 2.5 × ULN; If there is liver metastasis, ALT and AST should be ≤ 5 × ULN; Blood creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl) calculated according to the Cockcroft Gault formula ≥ 50 mL/min; International normalized ratio (INR) and activated partial thromboplastin time (aPTT): ≤ 1.5 × ULN (this standard is only applicable to patients who have not received anticoagulant therapy); Patients receiving anticoagulant therapy should ensure that the anticoagulant is within the required treatment range;

* Have not received systemic corticosteroid treatment within 4 weeks prior to treatment;
* Men with reproductive ability or women with the possibility of pregnancy must use highly effective contraceptive methods during the trial (such as oral contraceptives, intrauterine devices, abstinence control or barrier contraception combined with spermicides), and continue contraception for 12 months after the end of treatment;
* The subjects voluntarily joined the study, signed informed consent forms, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Previous treatment with anti-PD-1, anti-PD-L1, and anti-PD-L2, including adjuvant therapy phase;
* Individuals known to be allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components;
* Those who have received systemic chemotherapy, radiation therapy, or other anti-tumor treatments (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks before the start of treatment, or have not yet recovered from the previous toxicity (excluding 2nd degree hair loss and 1st degree neurotoxicity);
* Pregnant or lactating women;
* Positive HIV test result;
* Active hepatitis B or C patients HBsAg or HBcAb positive individuals were simultaneously detected with HBV DNA copy number positivity (quantitative detection limit is 500IU/ml, or reaching the copy number positivity value detected by the research center); Patients of this type must undergo HBV DNA testing during screening studies; Patients with positive HCV antibody test results are only eligible for this study if their HCV RNA PCR test results are negative;
* Have a clear history of active tuberculosis;
* Active autoimmune diseases that require systematic treatment within the past 2 years (such as the use of disease regulating drugs, corticosteroids, or immunosuppressive drugs), allowing for related alternative treatments (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for renal or pituitary dysfunction);
* Other serious and uncontrollable concomitant diseases that may affect the compliance of the scheme or interfere with the interpretation of the results, including active opportunistic infections or progressive (serious) infections, uncontrollable diabetes, cardiovascular diseases (Grade III or IV heart failure defined by the New York Heart Association classification, Grade II or above heart block, myocardial infarction, unstable arrhythmia or unstable angina pectoris in the past six months, cerebral infarction in three months, etc.) or lung diseases (interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm history);
* Previously received live vaccination within 4 weeks before the start of treatment;
* Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Significant surgical procedures (excluding diagnostic surgeries or TURBT) performed within the 4 weeks prior to the start of treatment;
* Individuals with a history of substance abuse and inability to quit, or those with a history of mental disorders;
* Large amounts of pleural or ascites accompanied by clinical symptoms or requiring symptomatic treatment;
* In the past 5 years, have had other malignant tumors that have not been cured, but do not include malignant tumors that have been clearly cured, or curable cancers such as basal or squamous cell carcinoma, localized low-risk prostate cancer, cervical in situ cancer, or breast in situ cancer; Note: Localized low-risk prostate cancer (defined as patients with stage ≤ T2b, Gleason score ≤ 7, and PSA ≤ 20ng/mL (as measured) at the time of prostate cancer diagnosis who have received curative treatment and have no biochemical recurrence of prostate-specific antigen (PSA) may participate in this study);
* Simultaneous presence of upper urinary tract urothelial carcinoma (renal pelvis, ureteral urothelial carcinoma);
* According to the researcher's perspective, there may be increased risks associated with participating in the study, or other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that may interfere with the interpretation of the research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-month Complete Response (3-month CR) | 3 months
  Three months after the start of treatment, if there is no visible tumor detected by imaging examination, the pathological evaluation of the tumor site obtained by diagnostic TURBT/cystoscopy is negative, and the urine cytology(for example, urine TCT) is negative, it is defined as CR. For the primary efficacy endpoint CR, the exact binomial distribution method will be used to provide point estimates, 95% confidence intervals, and p-values for testing response rates higher than the historical control (20%).

SECONDARY OUTCOMES:
6/12/24-month Complete Response (6/12/24-month CR) | 6/12/24 months
  The complete response rate (CR) after 6/12/24 months of treatment initiation is defined as the absence of visible tumors on imaging examinations, negative pathological evaluation of tumor site obtained by diagnostic TURBT/cystoscopy, and negative urine cytology( for example: urine TCT ) in subjects after treatment. For the primary efficacy endpoint CR, the exact binomial distribution method will be used to provide point estimates, 95% confidence intervals, and p-values for testing response rates higher than the historical control (20%).
Bladder Intact Event-Free Survival (BI-EFS) | 2 years
  Record the survival time of patients with preserved bladder function after treatment and no specific adverse events (such as tumor recurrence, metastasis, death, or the need for bladder resection). Provide Kaplan Meier (KM) curves and median estimates as appropriate.
Relapse-Free Survival (RFS) | 2 years
  During the treatment and follow-up period, the recurrence of previously disappeared tumors was suspected by urine cytology (such as tct), imaging (such as MRI) and confirmed by cystoscopy or pathology, which is defined as recurrence. If there is a recurrence, record the local recurrence time and distant recurrence time. For statistical analysis of results, provide Kaplan Meier (KM) curves and median estimates as appropriate
Cancer-Specific Survival (CSS) | 2 years
  From the first treatment (surgery, TURBT), record whether these patients died of bladder cancer (for example, due to tumor progression, metastasis or cancer related complications, such as renal failure or sepsis secondary to obstruction), and calculate the time. And exclude (non CSS events): death from unrelated conditions (such as myocardial infarction, stroke, trauma) or secondary primary cancer due to the following reasons (unless it is proved to be metastasis or recurrence of bladder cancer). Tumors are detected every 3/6 months through urine cytology (such as TCT), imaging (such as CT, MRI), and confirmed by cystoscopy or pathology.
Overall Survival (OS) | 2 years
  Starting from the first treatment (surgery, TURBT), record whether these patients have died. Tumors are detected every 3/6 months through urine cytology (such as TCT), imaging (such as CT, MRI), and confirmed through cystoscopy or pathology. OS =date of death - start date of treatment. For patients who were still alive or lost to follow-up at the last follow-up, the last follow-up date will be used as the cutoff. For statistical analysis of results, provide Kaplan Meier (KM) curves and median estimates as appropriate.
Adverse Event (AE) | 2 years
  During the study, adverse events will be monitored and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 guidelines. The efficacy evaluation of the subjects is confirmed by the researchers. After the end of treatment, outpatient or telephone follow-up will be conducted to investigate potential adverse events related to the study drug for at least 30 days after the last use of the subject's medication (serious adverse events potentially related to the study drug within 90 days after the last use of the subject's medication will be collected). For any AE, any severe AE, any grade 3-5 AE, any drug-related AE, any severe drug-related AE, any grade 3-5 drug-related AE, suspension of medication due to AE, discontinuation of medication due to AE, any immune related AE (irAE), mortality, and the incidence of specific AE, summary statistics will be provided in terms of quantity, percentage, and 95% confidence interval.
Biomarkers | 2 years
  Collect and detect the expression of relevant biomarkers (such as utDNA) in tumor tissue, urine, and blood at baseline, before each visit during treatment, and after completion of all treatments in the outpatient department. Perform sequencing to determine and analyze the correlation with therapeutic efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medecine, Shanghai, Shanghai Municipality, China